CLINICAL TRIAL: NCT02554006
Title: Predischarge Bundle for Patients in Dual Antiplatelet Therapy to Minimize the Negative Impact of Nuisance Bleedings on Quality of Life: a Randomized Controlled Trial.
Brief Title: Predischarge Bundle to Minimize Negative Impact on Quality of Life of Nuisance Bleedings
Acronym: BATMAN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital of Ferrara (Other)
Responsible Party: Principal Investigator, Gianluca Campo, interventional cardiologist and assistant professor, University Hospital of Ferrara
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 150595
Record Dates: First submitted 2015-09-17; First posted 2015-09-18 (Estimated); Last update posted 2018-05-02 (Actual); Status verified 2018-05

CONDITIONS: Myocardial Ischemia; Hemorrhage; Quality of Life; Platelet Aggregation Inhibitors
MeSH Terms: conditions — Myocardial Ischemia; Hemorrhage | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- good clinical practice (Other): all patients will receive education from physician regarding management of dual antiplatelet therapy as part of the routine discharge process
  Interventions: Behavioral: good clinical practice
- bundle group (Experimental): patients assigned to the bundle group will receive visits and materials as described by the protocol (counseling)
  Interventions: Behavioral: bundle group

INTERVENTIONS:
Behavioral: good clinical practice — education from physician regarding dual antiplatelet therapy as part of the routine discharge process
  Other Names: standard of care
  Arms: good clinical practice
Behavioral: bundle group — visits and materials describing advantages and side effects of dual antiplatelet therapy and their management
  Other Names: counseling regarding dual antiplatelet therapy management
  Arms: bundle group

SUMMARY:
A single-center, randomized trial of admitted patients with ischemic heart disease receiving percutaneous coronary intervention and stent implantation will be conducted at University Hospital of Ferrara. Patients will be randomized to either the control (standard care) or the bundle group in which patients will receive counseling regarding dual antiplatelet therapy management, advantages and side effects, screening for depression or anxiety, standardized education. The primary endpoint will be the difference in the quality of life as assessed by EQ-5D questionnaire.

DETAILED DESCRIPTION:
Recent studies suggest that bleeding complications have a strong influence on quality of life. During DAPT regimen bleeding complications occur from 5% to 15% of patients. Nuisance bleedings (BARC 1 bleeding) occur more frequently and show a strong influence on quality of life, depression, anxiety and compliance to the treatment.

The aim of the study is to establish if a specific counseling programme might minimize the negative quality of life impact of nuisance bleedings. A computer-generated list will be used to randomize patients in a 1:1 ratio, stratified by age, sex, renal failure and P2Y12 inhibitor, to either the bundle or the control group.

All patients randomized to the control group (standard of care) will receive education from physician regarding dual antiplatelet therapy (DAPT) as part of the routine discharge process.

All patients randomized to the bundle group will receive:

i) a 15-min visit by a member of the research team 24 h prior to the anticipated discharge day. During this visit, a core set of DAPT risks will be addressed. Advantages and side effects of DAPT will be described. The importance of compliance will be discussed. The correct management of side effects (especially BARC 1 bleedings) will be discussed.

ii) a 15-min visit by a member of the research team with a family member living near/with the patient. Advantages and side effects of DAPT will be described. The importance of compliance will be discussed. The correct management of side effects (especially BARC 1 bleedings) will be discussed.

iii) brochure describing advantages, side effects and management of dual antiplatelet therapy. Contemporaneously, the investigators of the study will contact directly by phone and/or mail the general practionnaire of the patient to describe and explain the same topics and the clinical problem of her patient.

iv) availability of phone number to discuss potential side effects of DAPT. In addition, the study coordinator of the study will contact two times by month the patient by phone to assess DAPT compliance and potential BARC 1 bleedings.

ELIGIBILITY:
Inclusion Criteria:

* signed written informed consent
* hospital admission for ischemic heart disease with clinical indication to coronary artery angiography
* percutaneous coronary intervention and drug eluting stent implantation
* indication to dual antiplatelet therapy for at least 6 months

Exclusion Criteria:

* oral anticoagulant therapy
* bleeding event in the 30 days before the enrolment
* planned surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 448 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2016-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
quality of life | 1 month
  quality of life assessment in each patient by EQ-5D questionnaire

SECONDARY OUTCOMES:
emergency room admission | 1 month
  number of access to emergency room service for bleeding
general practitioner visit | 1 month
  number of access to general practitioner for bleeding
dyspnea occurrence | 1 month
  number of patients suffering dyspnoea stratified according P2Y12 inhibitors
bleeding academic research consortium (BARC) 2-3 | 1 month
  occurrence of BARC 2-3 complications
bleeding academic research consortium (BARC) 1 | 1 month
  occurrence of BARC 1 complications

OTHER OUTCOMES:
ischemic adverse events | 1 year
  cumulative incidence of the following ischemic adverse events: cardiac death, myocardial infarction, transient ischemic attack/stroke
all-cause mortality | 1 year
  occurrence of all-cause death
BARC 1-3 | 1 year
  occurrence of BARC1-3 complications

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Ferrara, Cona, Ferrara, Italy

REFERENCES:
- [Result] Biscaglia S, Tonet E, Pavasini R, Serenelli M, Bugani G, Cimaglia P, Gallo F, Spitaleri G, Del Franco A, Aquila G, Vieceli Dalla Sega F, Tebaldi M, Tumscitz C, Ferrari R, Campo G. A counseling program on nuisance bleeding improves quality of life in patients on dual antiplatelet therapy: A randomized controlled trial. PLoS One. 2017 Aug 23;12(8):e0182124. doi: 10.1371/journal.pone.0182124. eCollection 2017. PMID 28832589